CLINICAL TRIAL: NCT01074021
Title: A Prospective,Randomized,Double-Blind,Controlled,Multicenter,Phase III Study of Nimotuzumab in Combination With Chemotherapy and Radiotherapy for Patients With Local Advanced Nasopharyngeal Cancer
Brief Title: Nimotuzumab in Combination With Chemoradiation for Nasopharyngeal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BT-CT-001
Record Dates: First submitted 2010-02-21; First posted 2010-02-24 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-08

CONDITIONS: Nasopharyngeal Cancer
Keywords: Nimotuzumab; Nasopharyngeal cancer; chemoradiation
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — nimotuzumab; Chemoradiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nimotuzumab plus chemoradiotherapy (Experimental)
  Interventions: Drug: Nimotuzumab
- placebo plus chemoradiotherapy (Placebo Comparator)
  Interventions: Drug: placebo plus chemoradiotherapy

INTERVENTIONS:
Drug: Nimotuzumab — Nimotuzumab:(200mg/w,weekly, 7-8 weeks, one week before radiotherapy)
  Radiotherapy:
  IMRT: Nasopharynx: GTV 66-78. 2Gy,CTV1 60-64Gy,CTV2 54-60Gy.30-34 times, 2.20-2.30Gy/time,once a day, 5 days/w, 6-7 weeks. Neck: lymph node positive, GTVn 60-70Gy, once a day, 5 days/w, 6-7weeks; lymph node negative, CTVn50-55Gy, once a day, 5 days/w, 6-7 weeks.
  CRT: Nasopharynx, 70-(76-80)Gy, 35-(38-40)times, 2Gy/time, once a day, 5 days/w, 6-8weeks. If disease residual when radiotherapy finished could increase the dose appropriate. Neck: lymph node positive, 64-70 Gy, 32-35 times, 2 Gy/time, once a day, 5 days/w, 6-7 weeks; lymph node negative, 50-56 Gy, 25-28 times,2 Gy/time, once a day, 5 days/w, 5-6weeks cisplatin
  Chemotherapy:
  Cisplatin (100 mg/m2,1 time/21d, 3 times，on days 2, 23, 44 during the radiotherapy)
  Arms: Nimotuzumab plus chemoradiotherapy
Drug: placebo plus chemoradiotherapy — Placebo treatment:4 bottles/w,weekly, 7-8 weeks, one week before radiotherapy
  Radiotherapy:
  IMRT: Nasopharynx: GTV 66-78. 2Gy,CTV1 60-64Gy,CTV2 54-60Gy.30-34 times, 2.20-2.30Gy/time,once a day, 5 days/w, 6-7 weeks. Neck: lymph node positive, GTVn 60-70Gy, once a day, 5 days/w, 6-7weeks; lymph node negative, CTVn50-55Gy, once a day, 5 days/w, 6-7 weeks.
  CRT: Nasopharynx, 70-(76-80)Gy, 35-(38-40)times, 2Gy/time, once a day, 5 days/w, 6-8weeks. If disease residual when radiotherapy finished could increase the dose appropriate. Neck: lymph node positive, 64-70 Gy, 32-35 times, 2 Gy/time, once a day, 5 days/w, 6-7 weeks; lymph node negative, 50-56 Gy, 25-28 times,2 Gy/time, once a day, 5 days/w, 5-6weeks cisplatin
  Chemotherapy: Cisplatin (100 mg/m2,1 time/21d, 3 times，on days 2, 23, 44 during the radiotherapy)
  Arms: placebo plus chemoradiotherapy

SUMMARY:
Nimotuzumab is an IgG1 humanized monoclonal antibody that recognized an epitope located in the extra cellular domain of the human epidermal growth factor receptor (EGFR). Clinical trials are ongoing globally to evaluate nimotuzumab in different indications. Nimotuzumab has been granted approval for use in squamous cell carcinoma of head and neck (SCCHN), glioma and nasopharyngeal cancer in different countries. The Clinical efficacy has been shown in adult with head and neck cancer. The study assessed the clinical efficacy, and safety of the combination of Nimotuzumab administered concomitantly with chemotherapy and radiotherapy in patients with advanced nasopharyngeal cancer.

DETAILED DESCRIPTION:
Patients with advanced nasopharyngeal cancer will be randomized to 2 arms. The patients in experimental arm will be treated with Nimotuzumab which will be used concurrently with radiotherapy and chemotherapy. The chemotherapy regimen were Cisplatin monotherapy. The active comparator arm will be administered chemotherapy and radiotherapy only. The dose and regimen were the same with experiment arm. The patients'hematopoietic , hepatic and renal function tests will be monitored weekly, a physical exam and reassessment of the tumor will be performed at the first and the fourth month, and followup every six months to evaluate the survival index in three years after the study.

ELIGIBILITY:
Inclusion Criteria:

* Joined the study voluntary and signed informed consent form
* Age 18-70，both genders.
* Nasopharyngeal cancer was confirmed by pathology.
* Nasopharyngeal cancer 2008 Stages: Ⅲ/Ⅳa.
* Primary lesions can measurable.
* Karnofsky Performance Scale >70.
* Life expectancy of more than 6 months.
* Use of an effective contraceptive method for women when there is a risk of pregnancy during the study.
* Haemoglobin≥100g/L ,WBC ≥4×109/L, platelet count≥100×109/L
* Hepatic function:ALAT、ASAT< 1.5 x ULN, TBIL< 1.5 x ULN
* Renal function: Creatinine < 1.5 x ULN

Exclusion Criteria:

* Evidence of distant metastasis
* Primary lesions or lymph node have been operated (except of operation for biopsy)
* Previous radiotherapy
* Received other anti EGFR monoclonal antibody treatment
* Previous chemotherapy or immunization therapy
* Other malignant tumor (except of Non-melanoma Skin Cancer or carcinoma in situ of cervix)
* Participation in other interventional clinical trials within 1 month
* Peripheral neuropathy is more than I stage
* Pregnant or breast-feeding women and women who refused to take contraceptive method
* History of serious allergic or allergy
* History of Serious lung or heart disease
* Refused or can't signed informed consent form
* Drug abuse or alcohol addiction
* Personality or psychiatric disease, and persons without capacity for civil conduct or persons with limited capacity for civil conduct

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2009-10; Primary Completion 2016-05 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
To determine the local-regional control rates of the disease in the advanced nasopharyngeal cancer patients subject to the treatment with Nimotuzumab in combination with chemoradiation | 3 months after the Nimotuzumab treatment finished
To determine the safety of the treatment with Nimotuzumab in combination with chemoradiation | within study period

SECONDARY OUTCOMES:
To determine the Disease-free survival、Tumor control probability、Distant recurrence rate in the patients subject to the treatment at years 1,2,3 | 3 year
To determine the Progression free suivival、Diease free survival、Overall survival in the patients subject to the treatment | 3 years

CONTACTS AND LOCATIONS:
Locations (24):
- China (24):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Xiamen First Hospital, Xiamen, Fujian
  - The Affiliated Cancer Hospital of Guangzhou Medical Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Affiliated Tumor Hospital of Guangxi Medical University, Xining Shequ, Guangxi
  - The Fourth Hebei Province Hospital, Shijiazhuang, Hebei
  - The Affiliated Cancer Hospital of Haerbin Medical University, Haerbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Province Caner Hospital, Wuhan, Hubei
  - Wuhan Union Hospital, Wuhan, Hubei
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Province Cancer Hospital, Shenyang, Liaoning
  - Shandong Caner Hospital, Jinan, Shandong
  - Sichuan Province Cancer Hospital, Chengdu, Sichuan
  - West China School of Medicine/West China Hospital of Sichuan University (WCSM/WCH), Chengdu, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Cancer Institute & Hospital.Chinese Academy of Medical Sciences, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - The General Hospital of the People's Liberation Army, Beijing
  - The Affiliated Renji Hosptial of ShanghaiJiao Tong University, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Cancer Hospital, Tianjin